CLINICAL TRIAL: NCT02279654
Title: A Post-authorization, Non-interventional, Safety Study Study of Patients With Myelodysplastic Syndromes (MDS) Treated With Lenalidomide.
Brief Title: Non-interventional Study of Lenalidomide in the Clinical Routine Treatment of TD Patients With IPSS Low or Int-1 MDS and Isolated Del(5q)
Acronym: PASS MDS del5q
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-5013-MDS-010
Record Dates: First submitted 2014-10-21; First posted 2014-10-31 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Myelodysplastic Syndrome
Keywords: Lenalidomide; Revlimid; Transfusion-dependent; international Prognostic Scoring System (IPSS) low; Intermediate-1-risk; MDS; Isolated del(5q); Prospective; Non-interventional; Post-authorization safety study (PASS); Disease registry
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lenalidomide Population: Patients with transfusion-dependent, low- or intermediate (int)-1risk MDS and isolated del (5q) who receive at least 1 dose of lenalidomide after 15th June 2007 and have been followed up for on the registry for 3 years or until death/consent withdrawal
  Interventions: Drug: Lenalidomide
- Background Population: All MDS patients who have been diagnosed on 15th June 2007 or later, have never been exposed to lenalidomide and have been followed up on the registry for 3 years or until death/consent withdrawal
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide as prescribed in routine clinical practice for low to intermediate-1 risk MDS
  Other Names: Revlimid; CC-5013

SUMMARY:
This registry is a prospective, non-interventional, post authorisation safety study for patients diagnosed with Transfusion Dependent, IPSS low or intermediate-1-Risk Myelodysplastic Syndrome (MDS), associated to a single abnormality of the chromosome 5 [del(5q)].

The purpose of this study is to collect additional data about the safety of an oral drug (lenalidomide, Revlimid®) that may have been prescribed to relieve anemia and decrease the need of blood transfusions. However, also patients affected by the MDS del(5q) who receive other treatments different from lenalidomide can be included in this study, if they agree.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥ 18 years old at the time of signing the Informed consent form (ICF)
* Are transfusion dependent or have an history of transfusion dependence; for the purpose of the current Myelodysplastic syndromes (MDS) Post-authorization safety study (PASS), transfusion-dependence is defined as requiring ≥2 RBC units over an 8 week period prior to the date of signature on the ICF (due to MDS-related causes and not because of hemorrhage, trauma, or other acute cause)
* Are on active treatment with lenalidomide (Lenalidomide Cohort) or have never been exposed to lenalidomide at the time of signing the ICF (Background Cohort)
* Have confirmed diagnosis of IPSS low or intermediate-1-risk MDS with isolated del (5q) (with morphological and cytogenetic information) diagnosed on 15 June 2007 (date of Revlimid first approved in Europe) or later

Exclusion Criteria:

* Refuse to participate in the Myelodysplastic syndromes (MDS) Post-authorization safety study (PASS),
* Are currently participating in an interventional therapeutic clinical trial for MDS (except for erythropoiesis-stimulating agents [ESAs] and granulocyte colonystimulating growth factors)
* Receive any investigational agent the time of signing the ICF
* Have previously been treated with lenalidomide and are no longer on active treatment with lenalidomide at the time of signing the ICF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received at least 1 dose of any treatment or treatment modality after the patient signs the informed consent form
  * Lenalidomide cohort: All patients treated with lenalidomide
  * Background cohort: All patients treated with therapeutic modalities other than lenalidomide
  For each population 3 datasets will be described and will form the basis of subsequent analyses:
  * A baseline demographic dataset ("population dataset")
  * An exposure dataset
  * An outcome dataset
Sampling Method: Non-Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Ascertain the Disease Progression to AML (through calculation of product limit estimators and incidence rates) for those with transfusion dependent Low to Intermediate 1 risk MDS del 5 q and have been treated with Revlimid | Up to 3 years
  Incidence, as well as the attributable risk (AR) and AR percent (%). Progressive Disease criteria includes increasing monoclonal paraprotein levels, bone marrow findings, worsening lytic bone disease, progressively enlarging extramedullary plasmacytomas, or hypercalcemia.
Overall Survival for patients with transfusion-dependent low to intermediate 1 risk MDS and isolated del (5q) and who have been treated with Lenalidomide | Up to 3 years
  Number of MDS participants who survive

SECONDARY OUTCOMES:
Overall Survival for patients with transfusion-dependent low to intermediate 1 risk MDS and isolated del (5q) and who have been treated with Lenalidomide | Up to 3 years
  Number of MDS participants who survive who have never been treated with Lenalidomide
Adverse Events | Up to 3 years
  Type, frequency, severity of advere events and relationship of adverse events to Lenalidomide. An adverse ecent is defined as any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment, ie, any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product whether or not considered related to the medicinal product
Evaluate risk factors associated with progression of AML | Up to 3 years
  Employ Cox proportional hazards models among MDS patients included in the primary population who have been treated with lenalidomide
Clinical practice | Up to 3 years
  Provide insight into treatment regimens and therapy sequence in clinical practice as they relate to clinical outcomes (response, overall survival, progression-free survival) in patients in MDS participants

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (148):
- United States (13):
  - Local Institution - 0001, Centre City, New Jersey
  - Local Institution - 0002, Centre City, New Jersey
  - Local Institution - Belgium, No City Provided, New Jersey
  - Local Institution - Denmark, No City Provided, New Jersey
  - Local Institution - France, No City Provided, New Jersey
  - Local Institution - Germany, No City Provided, New Jersey
  - Local Institution - Greece, No City Provided, New Jersey
  - Local Institution - Italy, No City Provided, New Jersey
  - Local Institution - Luxembourg, No City Provided, New Jersey
  - Local Institution - Norway, No City Provided, New Jersey
  - Local Institution - Spain, No City Provided, New Jersey
  - Local Institution - Sweden, No City Provided, New Jersey
  - Local Institution - UK, No City Provided, New Jersey
- Belgium (7):
  - AZ Klina, Brasschaat
  - AZ Sint Jan, Bruges
  - GHdCharleroi, Charleroi
  - Jessa Ziekenhuis, Hasselt
  - CHR Citadelle, Liège
  - CHU Vésale, Montigny-le-Tilleul
  - Clinique Saint-Pierre Ottignie, Ottignies
- Denmark (5):
  - Aalborg Sygehus, Dept of Hematology, Aalborg
  - Århus University Hospital, Aarhus
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense
  - Rokslide Hospital, Roskilde
- France (17):
  - Hopital de L'archet I, Nice, Alpes-Maritimes
  - Institut Paoli Calmettes, Marseille, Bouches-du-Rhône
  - CHU Haut-Lévêque, Pessac, Gironde
  - CHU Hôtel Dieu, Nantes, Loire-Atlantique
  - CHU Hôtel Dieu, Angers
  - Centre Hospitalier D'Avignon - Hopital Henri Duffaut, Avignon
  - CH Chalon/Saone William Morey, Chalon-sur-Saône
  - CHU Grenoble, La Tronche
  - CHRU De Lille - Hôpital Claude - Rue Michel Polonovski, Lille
  - Centre Hospitalier Universitaire De Limoges - Hopital Dupuyt, Limoges
  - CHU Hôtel Dieu - Place A Ricordeau, Nantes
  - Hôpital St Louis, Paris
  - Centre Hospitalier Lyon-SUD [U, Pierre-Bénite
  - Hopital de Hautepierre CHRU de Strasbourg, Strasbourg
  - Hopital Purpan-Place du Dr. Baylac, Toulouse
  - CHU Bretonneau, Tours
  - CHU Nancy Brabois Adultes - 58 Allee dy morvan, Vandœuvre-lès-Nancy
- Germany (26):
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld
  - Hämatologie und Onkologie, Klinikum Chemnitz gGmbH International Patient Center, Chemnitz
  - Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Universitätsklinik Carl-Gustav, Dresden
  - HELIOS St. Johannes Klinik, Duisburg
  - Uniklinikum Düsseldorf, Klinik für Hämatologie, Onkologie und Klinische Immunologie, Düsseldorf
  - Marien Hospital Düsseldorf, Düsseldorf
  - St Antonius Hospital (SAH), Eschweiler
  - Kreiskrankenhaus St. Elisabeth - Von Werth-Str., Grevenbroich
  - Praxis, Onkologische Schwerpunktpraxis Dres. Verpoort, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Institut für Versorgungsforschung in der Onkologie, Koblenz
  - InVO Institut fur Versorgungsforschung, Koblenz
  - Gemeinschaftspraxis fur Hamatologie und Onkologie, Onkologisches zentrum Lebach, Lebach
  - Abteilung Hämatologie, Internistische Onkologie, Universitatklinikum Leipzig, Leipzig
  - III. Medizinische Klinik, Hämatologie und internistische Onkologie , Univesitatsmedizin Mannheim, Mannheim
  - Gesellschaft für Medizinische, Mönchengladbach
  - MLL Münchner Leukämielabor GmbH, München
  - III. Medizinische Klinik, Klinikum rechts der Isar der Technischen Universität München, München
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Innere Medizin II - Onkologie, Hämatologie, Univesitatklinikum Tubingen, Tübingen
  - Klinik für Innere Medizin III, Ulm
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Westerstede
  - Rems-Murr-Klinikum Winnenden, Winnenden
  - Universitätsklinikum Würzburg, Würzburg
  - ZENTRUM FÜR INNERE MEDIZIN, Universitatklinikum Wurzburg, Würzburg
- Greece (9):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - General Hospital of Athens - LAIKO, Athens
  - University General Hospital, Athens
  - Georgios Gennimatos General Hospital, Athens
  - University Hospital Of Herakli, Herakleion - Crete
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - University General Hospital of Patras, Pátrai
  - G. Papanikolaou General Hospital, Thessaloniki
- Italy (22):
  - Irccs Crob, Rionero in Vulture, Potenza
  - Ospedale di Castelfranco Venet, Castelfranco Veneto, Treviso
  - AOU Ospedali Riuniti Umberto I G.M. Lancisi G. Salesi, Ancona
  - U.O Ematologia con Trapianto, Bari
  - Azienda Ospedaliera Papa Giovanni XX111 Piazza OMS, Bergamo
  - Policlinico S.Orsola Malpighi, AOU di Bologna, Bologna
  - AO Spedali Civili di Brescia, Brescia
  - Policlinico di Catania, Catania
  - AOU Careggi, Florence
  - U.O .C di Oncoematologia, Mirano
  - Ospedale S. Luigi Gonzaga, Orbassano
  - Azienda ospedaliero-universita, Parma
  - Azienda Ospedaliera di Perugia, Perugia
  - Ospedale Civile Santo Spirito, Pescara
  - Arcispedale S.Maria Nuova, Reggio Emilia
  - U.O Ematologia Azienda Ospedaliera, Regio Calabria
  - Univesita La Sapienza, Roma
  - AOU Policlinico Tor Vergata, Università Roma Tor Vergata, Roma
  - Presidio Ospedaliero "A. Torto, Salerno
  - Azienda Ospedaliera Universitaria di Sassari, Sassari
  - A.O. Citta' della Salute e del, Torino
  - Policlinico "G.B. Rossi" Verona, Veneto
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Haukeland Sykehus, Bergen, Norway
- Spain (29):
  - Hospital Universitario de Gran Canaria Servicio de Hematología y, Las Palmas de Gran Canaria, Canary Islands
  - H.U.Marq.Valdecilla, Hospital Universitario Marqués de Valdecilla. Hematología, Santander, Cantabria
  - Hospital costa del sol, Marbella, Málaga
  - H.U. Ribera de Alzira, Alzira
  - Hospital de Cruces, Barakaldo
  - Hospital del Mar,Hematologia Hemotheropia, Barcelona
  - H. Clinic de Barcelona, Barcelona
  - Pauc Tauli, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Instit Catalia D'Oncologia, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital Josep Trueta (ICO Girona), Girona
  - Hospital Virgen de Las Nieves, Granada
  - Department of Hematology, Hospital Duran i Reynals, LLobregat
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hopsital Clinico San Carlos, Madrid
  - Hospital Universitario fundacion Jiminez Diaz, Madrid
  - Hospital Universitario 12 de Octobre, Madrid
  - Hospital Universitario La Paz, Madrid
  - H Universitario Puera de Hierro, Madrid
  - Hospital Son Espaces, Mallorca
  - Hospital Universitario central de Asturias, Oviedo
  - Univesity Hospital de Salamanca, Salamenca
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Virgen Macarena, Seville
  - Hospital Virgen del Rocio, Seville
  - Hopsital Nuestra Senora de Valme, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospiral Universitario de la Fe, Valencia
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Länssjukhuset Kalmar, Kalmar
  - Lund University Hospital - Lasarettsgatan 23, Lund
  - Karolinska University Hopsital, Stockholm
- United Kingdom (14):
  - Maidstone Hospital, Maidstone, Kent
  - Aberdeen Royal Infirmary - Foresterhill Road, Aberdeen
  - Queen Elizabeth Hospital, Birmingham
  - Pilgrim Hospital, Boston
  - Monkton, Wishaw and Hairmyres Hospitals, East Kilbride
  - Broomfield Hospital - Mid-Essex Hospitals NHS Trust, Essex
  - Basildon and Thurrock Hospitals, Essex
  - Northwick Park Hospital, Harrow
  - Lincoln county Hospital, Lincoln
  - Aintree Hospital - Longmoor Lane, Liverpool
  - University Hospital South Manc, Manchester
  - Royal Oldham Hospital, Oldham
  - Radcliffe Hospitals and University - Headley Way, Headington, Oxford
  - Great Western Hospital, Swindon